CLINICAL TRIAL: NCT02045784
Title: Establishing the Iodine Requirement in Infancy: a Double-blind Dose-response, Cross-over Balance Study
Brief Title: Establishing the Iodine Requirement in Infancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: North-West University, South Africa (Other)
Responsible Party: Principal Investigator, Maria Andersson, Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 2013-N-21
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Focus: Establish the Iodine Requirement During Infancy
MeSH Terms: interventions — Infant Formula; Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infant formula milk 60 µg iodine/day (Experimental): Infant formula containing 57 µg/100 g powder, providing approximately 60 µg iodine/day (i.e. 55% of the current AI). Unrestricted consumption during 11 days.
  Interventions: Dietary Supplement: Infant formula
- Infant formula milk 110 µg iodine/day (Experimental): Infant formula containing 92 µg/100 g powder, providing approximately 110 µg iodine/day (i.e. 100% of the current AI). Unrestricted consumption during 11 days.
  Interventions: Dietary Supplement: Infant formula
- Infant formula 220 µg iodine/day (Experimental): Infant formula containing 217 µg/100 g powder, providing approximately 220 µg iodine/day (i.e. 200% of the current AI). Unrestricted consumption during 11 days.
  Interventions: Dietary Supplement: Infant formula
- Breast milk (Other): Unrestricted consumption during 4 days
  Interventions: Other: Breast milk

INTERVENTIONS:
Dietary Supplement: Infant formula — To establish dose-response relationships, formula-fed infants will be randomly allocated to three 11-day cross-over periods of exclusive consumption of infant formula providing different amounts of iodine. All iodine levels are within the required iodine levels for infant formula following the regulations of the United States, the European Union, Switzerland and New Zealand.
  Arms: Infant formula 220 µg iodine/day; Infant formula milk 110 µg iodine/day; Infant formula milk 60 µg iodine/day
Other: Breast milk — Unlimited breast feeding
  Arms: Breast milk

SUMMARY:
The objective of this study is to define the amount of dietary iodine needed per day during the first six months of life. The hypothesis is that the current recommended iodine intake in infants is set too high.

DETAILED DESCRIPTION:
Iodine is an essential trace element for human health and an integral component of the thyroid hormones. Thyroid hormones regulate normal growth and development, particularly of the brain. Iodine deficiency results in low levels of thyroid hormones that can impair brain development and lower intelligence. Infants have only small iodine stores at birth and are entirely dependent on iodine provided by breast milk or infant formula. However, the exact amount of daily iodine that infants need for healthy development is poorly understood and there is insufficient data to define an Estimated Average Requirement (EAR) for this age group.

The current recommendation for dietary iodine intake for 0-6 month (mo) old infants of 110 µg/day is only an adequate intake (AI), in the absence of an EAR. This AI is based on the iodine intake in breast fed infants from breast milk iodine concentration (BMIC) measured in U.S. women during a period when overall iodine intakes in the U.S. population were excessive. The AI sharply disagrees with the current WHO recommendation for assessment of infant iodine nutrition based on excretion of iodine in the urine. The discrepancy makes assessment and monitoring of iodine status at this age problematic and has led to major confusion on how to interpret adequate iodine intake and optimal iodine status.

The objective of this study is to measure the daily iodine retention from dietary iodine and define the physiological iodine requirement (the EAR) during the first six months of life. The study hypothesis is that the AI is set too high and its use in assessing iodine intake and status overestimates the prevalence of iodine deficiency in infants.

The study will be a metabolic balance study of breast milk consumption and three dose-response cross-over arms of iodine enriched infant formula milk in 60 healthy 2-3 mo old infants (30 breast fed and 30 formula fed). Breast fed infants will be exclusively and unrestrictedly breast fed by the mother and the breast milk consumption will be monitored for 4 days by weighing the infants before and after each feeding session. Formula fed infants will be randomly allocated to three 11 days cross-over periods of exclusive consumption of infant formula milks (IFM) providing 60 µg I/day, 110 µg I/day and 220 µg I/day. The iodine intake will be monitored by recording the amount of infant formula milk fed to the infants. The iodine excretion will be measured from complete collections of urine and feces for a 4-day period for each arm. The iodine retention will be calculated from the difference between measured iodine intake and excretion. Analytical determination of the iodine content in biological samples will be done by mass spectrometry after digestion and iodine extraction. The sample size is based on an estimated dose-response of the different levels of dietary iodine on iodine excretion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mother/infant pairs (considering the following criteria: normal thyroid function, adequate iron status, no apparent infection)
* Full term birth (in week 38 to 42), birth weight >2 500 g, singleton birth
* No known family history of thyroid disease
* Infant does not have persistent stomach and/or intestine symptoms
* Mother did not use: a) X-ray or CT contrast agent (both may contain iodine); b) iodine containing medication within the last year
* Formula fed infants study arm: Infant is fully formula fed and was already formula fed prior to the study
* Formula fed infants study arm: Infant was fed with formula based on cow's milk protein prior to the study
* Formula fed infants study arm: Infant shows no signs of cow's milk allergy
* Breast fed infants study arm: Infant is fully breast fed and was fully breast fed prior to the study

Ages: 5 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Iodine retention | 4 days
  The amount of iodine retained will be calculated as the difference between measured iodine intake and measured iodine excretion

CONTACTS AND LOCATIONS:
Overall Officials: Maria Andersson, PhD, Principal Investigator — ETH Zurich
Locations (2):
- North-West University South Africa, Potchefstroom, South Africa
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Dold S, Zimmermann MB, Baumgartner J, Davaz T, Galetti V, Braegger C, Andersson M. A dose-response crossover iodine balance study to determine iodine requirements in early infancy. Am J Clin Nutr. 2016 Sep;104(3):620-8. doi: 10.3945/ajcn.116.134049. Epub 2016 Jul 27. PMID 27465383